CLINICAL TRIAL: NCT06616610
Title: Single-Button Mobility Platform's Effect on Reaction Time and Keystroke Accuracy in Children with Cerebral Palsy: a Pilot Study
Brief Title: Single-Button Mobility Platform's Effect on Reaction Time and Keystroke Accuracy in Children with Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Félix Biscarri Triviño, Head of research group, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PEIBA_0669-N-22
Record Dates: First submitted 2024-09-20; First posted 2024-09-27 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy Infantile
Keywords: Cerebral Palsy; Children; Reaction Time; mobility platform; cognitive development; GMFCS levels IV-V; motor skills
MeSH Terms: conditions — Cerebral Palsy | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Experimental Arm (Experimental): Participants included in arms are children with the following inclusion criteria:
  * Diagnosed with cerebral palsy
  * Classified as GMFCS level IV or higher, indicating an inability to walk or operate a powered wheelchair.
  * Under 12 years old.
  * Must be affiliated to a center whose facilities guarantee a proper navigation experience
  The participants will be randomly assigned to two equal-sized arms: the control arm, in which participants will continue with the traditional therapy, and the experimental arm, where the children will use the platform.
  The experimental arm receives an intervention (procedure) that is a focus of the study. It aims to analyze the impact of a single-button-operated mobility platform on reaction times and keypress patterns in children with severe disabilities.
  Interventions: Behavioral: Intervention with the Mobility Platform
- The Control Arm (Active Comparator): Participants included in arms are children with the following inclusion criteria: - Diagnosed with cerebral palsy - Classified as GMFCS level IV or higher, indicating an inability to walk or operate a powered wheelchair. - Under 12 years old. - Must be affiliated to a center whose facilities guarantee a proper navigation experience The participants will be randomly assigned to two equal-sized arms: the control arm, in which participants will continue with the traditional therapy, and the experimental arm, where the children will use the platform. The control arm participants continue with their regular therapy. Regular cause-effect therapies use an animated cartoon video that frequently pauses so that the children have to press an adapted button to continue watching it.
  Interventions: Behavioral: Intervention with Traditional Therapy

INTERVENTIONS:
Behavioral: Intervention with the Mobility Platform — The experimental arm receives the Intervention with Mobility Platform that is a focus of the study. It aims to analyze the impact of a single-button-operated mobility platform on reaction times and keypress patterns in children with severe disabilities.
  Arms: The Experimental Arm
Behavioral: Intervention with Traditional Therapy — The traditional cause-effect therapies use an animated cartoon video that frequently pauses so that the children have to press an adapted button to continue watching it.
  Arms: The Control Arm

SUMMARY:
The goal of this clinical trial is to determine whether the use of a mobility platform can improve response time in children with cerebral palsy.

The primary question it seeks to answer is: Can the use of a mobility platform enhance cognitive development in children with severe disabilities?

Children are randomly assigned to two equal-sized groups: the control group, where participants will continue with their standard therapy, and the intervention group, where participants will use the mobility platform. Researchers will compare outcomes between the two groups.

Participants in the control group will engage in a traditional cause-and-effect therapy, using a video that frequently pauses, requiring them to press an adapted button to continue watching. Participants in the intervention group will use the mobility platform during their sessions. Movement begins when the participant presses the adapted button, and the platform advances, adjusting its direction using sensors to detect obstacles. Once the preset time limit is reached, the platform stops, and the child must press the button again to resume movement. This stop-start process mirrors the cause-and-effect training in the control group.

DETAILED DESCRIPTION:
The experimental timeline includes eight weekly sessions, each lasting 30 minutes. Initially, therapists will receive an explanation on how to use the platform and the accompanying configuration application. They will familiarize themselves with it a couple of weeks before the experiment begins. During the sessions, children in the experimental group will use the platform, while those in the control group will continue receiving their traditional therapy.

Researchers will pre-adjust the children's interactions to match the platform variables, allowing for meaningful comparisons. Therapists will assess changes in the children's mood or emotional state during each session. To do this, they will calculate the differences between the SAM (Self-Assessment Manikin) tests conducted at the beginning and end of each session. A positive difference in valence indicates an improvement in the participant's happiness or positive emotions during the session. Similarly, positive changes in arousal reflect increased calmness or reduced excitation. A seven-item Likert scale will be used for measurement. For instance, if there is a positive change of seven points in valence during a session, the participant moves from a very sad state to a very happy one.

To minimize bias in conducting the experiment and evaluating SAM tests, therapists will be randomly assigned to either the control or intervention groups for each session, while ensuring an equal number of sessions conducted by each therapist. As a result, each therapist will conduct four sessions with the experimental group and four with the control group, with random session assignments.

The dependent variables include reaction time (RT) and the number of incorrect selections (NIS). The mean and standard deviation of these dependent variables allow for the following statistical analyses: Kruskal-Wallis Test: This will be used to compare the dependent variables across groups. SAM Test: It will score the statistically significant differences between the experimental and control groups, with the level of significance set at 5% (p = 0.05). Pearson Regression Analysis: This will identify trends in the dependent variables over time.

The registration procedure is as follows: Variables are collected, transmitted, and stored in a database on a cellphone for later analysis. To achieve this, the investigators used an Open Source Frontend SDK , which enables the deployment of hybrid mobile applications based on web development tools such as HTML, CSS, and JavaScript. The apps run in a browser shell. Several Capacitor plugins were used to manage the database and Bluetooth connectivity, which are essential for data storage and communication. The application interface includes buttons for therapists to enable/disable Bluetooth connections, start/stop recording, and a panic button to halt the platform and abort the experiment. Additionally, users can select their username and group name. Control group therapy involves the use of educational resources that require children to press a button repeatedly. For this group, the investigators chose fairy tale or cartoon videos from YouTube. The specific videos will be tailored to the user's preferences. These videos pause intermittently and require the child to perform an action to resume playback. A microcontroller is used to record time intervals and host an application that detects the child's keystrokes. This data is transmitted via Bluetooth to the same mobile application used for the mobility platform, ensuring synchronization between the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cerebral palsy
* Classified as GMFCS level IV or higher, indicating an inability to walk or operate a powered wheelchair.
* Under 12 years old.
* Must be affiliated to a center whose facilities guarantee a proper navigation experience

Exclusion Criteria:

- Inability to act on an actuator (Start button)

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Reaction time (RT) | From enrollment to the end of treatment at 8 weeks
  In the intervention group, RT measures the time elapsed between the platform stopping and the user pressing the button to initiate a new navigation period.
  In the control group, RT measures the time elapsed between the video pausing and the user pressing the button to continue watching it
Number of incorrect selections (NIS) | From enrollment to the end of treatment at 8 weeks
  NIS represents the number of additional button presses recorded while the Platform is in motion and serves validation purposes. A high value of this variable, consistently maintained over time, suggests that the user is not performing the cause-effect experiment effectively.

SECONDARY OUTCOMES:
The Self-Assessment Manikin (SAM) test | From enrollment to the end of treatment at 8 weeks
  The Self-Assessment Manikin (SAM) test is used to assess the emotional changes in children during the experiment. It comprises a 7-level Likert scale (the scale ranges from 1 to 7) associated with a set of faces displaying various degrees of valence and arousal.
  Valence reflects how pleasant or unpleasant an emotion. A score of 1 represents the most unpleasant emotion, while a score of 7 represents the most pleasant emotion.
  Arousal refers to the level of physiological and psychological activation or intensity of an emotional experience. A score of 1 indicates low arousal (low physiological and psychological activation), and a score of 7 indicates high arousal (high activation).
  Thus, higher scores mean more positive valence (pleasant emotion) and higher arousal (greater intensity).

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Molina Cantero, PhD, Principal Investigator — University of Seville, Seville, Andalucia, Spain
Locations (1):
- University of Seville, Seville, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From november 2024
Access Criteria: Everyone will be able to access all the IPD and all the supporting information. It will be available on It will be available on the Research Data Repository of the University of Seville (IdUS). IdUS is part of the digital infrastructure for open science and offers University of Seville authors a platform to deposit their publications in open access and their research data.
URL: https://idus.us.es/

REFERENCES:
- See also: The Self-Assessment Manikin (SAM) is a non-verbal tool used to measure emotional responses across three dimensions: valence (pleasure), arousal, and dominance. — https://www.millisecond.com/download/library/selfassessmentmanikin
- Available data/document: Individual Participant Data Set — https://idus.us.es/ — The idUS repository is part of the digital infrastructures for open science guaranteed by the National Strategy for Open Science (ENCA). It allows authors from the University of Seville (US) to deposit their publications in open access and manage their research data according to FAIR principles (Findable, Accessible, Interoperable, and Reusable).